CLINICAL TRIAL: NCT01997762
Title: Can Resveratrol Improve Insulin Sensitivity and Preserve Beta Cell Function Following Gestational Diabetes?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Institute of Child Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B2013:151
Record Dates: First submitted 2013-11-13; First posted 2013-11-28 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2013-11

CONDITIONS: Gestational Diabetes
Keywords: resveratrol,; gestational diabetes,; beta cell function; history
MeSH Terms: conditions — Diabetes, Gestational | interventions — Resveratrol; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Corn starch capsules, 1 capsule twice a day for 3 months
  Interventions: Dietary Supplement: Placebo
- Resveratrol (Experimental): Resveratrol capsules, 250 mg twice a day for 3 months
  Interventions: Dietary Supplement: Resveratrol

INTERVENTIONS:
Dietary Supplement: Resveratrol — gel-coated capsules to be taken twice a day; one with breakfast and dinner
  Other Names: All Natural Resveratrol 98% Super Strength
  Arms: Resveratrol
Dietary Supplement: Placebo
  Other Names: Corn starch capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if resveratrol supplementation preserves beta cell function and insulin sensitivity in post-partum women following a first diagnosis of gestational diabetes. We hypothesize that daily supplementation with resveratrol will preserve beta cell function and insulin sensitivity.

DETAILED DESCRIPTION:
Our primary aim is to perform a randomized controlled trial of resveratrol for the improvement of insulin sensitivity and the preservation of beta cell function in post-partum women following a first diagnosis of gestational diabetes. Our long-term goal is to test resveratrol for the secondary prevention of gestational diabetes and type 2 diabetes. We have developed six conditions that should be satisfied by the study to justify project expansion. Therefore, we will be testing hypotheses and computing estimates for the following six outcomes: (1) recruitment numbers, (2) adherence to study treatment, (3) adherence to study visits, (4) insulin sensitivity measured at 12 months post-partum, (5) beta cell function measured at 12 months post-partum, and (6) adverse events.

The study is a single-site, parallel, double-blind, randomized, placebo-controlled trial. The study population consists of women recruited during pregnancy who had a confirmed first diagnosis of gestational diabetes, who do not have either diabetes or pre-diabetes when re-tested 3 months post-partum, and who have stopped breastfeeding by 9 months post-partum. They study intervention is resveratrol (or identical placebo) twice daily for a total of 12 weeks from 9 months to 12 months post-partum. Our planned sample size is 112 women based on the hypothesis testing and estimation considerations for the six above-mentioned outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (18 years of age or older) 3 months post-partum with a recent history of first diagnosis of gestational diabetes.
* Willingness to provide informed consent 3 months post-partum.

Exclusion Criteria:

* Abnormal glucose tolerance or type 2 diabetes recorded at 3 months post-partum.
* Breastfeeding beyond 9 months post-partum.
* Intention to consume resveratrol open label.
* Intention to drink red wine (more than 4 glasses per week) or eat foods high in resveratrol (grapes, grape juice, peanuts, peanut products).
* Unwillingness to use two approved types of contraception until one year post-partum and unwillingness to undergo pregnancy test at randomization.
* Twin pregnancy.
* Consuming medications with a risk of interaction with resveratrol.
* Liver disease.
* Unlikely to be able to comply with study follow-up as judged by social (e.g. transient, not permanent residents, etc.) or geographical considerations.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in beta cell function | baseline and 3 months after intervention
  Beta cell function will be assessed by calculating the Insulin Secretion Sensitivity Index-2, a ratio of the area under the curve (AUC) for glucose and the AUC for insulin after an oral glucose tolerance test.

SECONDARY OUTCOMES:
recruitment rates | recruitment rates will be followed throughout the recruitment phase, which is expected to take 2 years maximum
treatment adherence | 3 months after intervention
Change in insulin sensitivity | baseline and 3 months after intervention
  Insulin sensitivity will be assessed by calculating the homeostasis model of assessment of insulin resistance (HOMA-IR).

OTHER OUTCOMES:
change in liver function | baseline and 3 months after intervention
  liver function will be assessed by measuring plasma concentrations of alanine aminotransferase, aspartate aminotransferase, gamma glutamyltransferase, total bilirubin and conjugated bilirubin.
change in C-reactive protein | baseline and 3 months after intervention
change in glycated hemoglobin | baseline and 3 months after intervention
change in serum lipids | baseline and 3 months after intervention
change in plasma levels of resveratrol and resveratrol metabolites | baseline and 3 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Shayne P Taback, MD, Principal Investigator — University of Manitoba
Locations (1):
- Manitoba Institute of Child Health, Winnipeg, Manitoba, Canada